CLINICAL TRIAL: NCT05023525
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, and Pharmacokinetics of Single Ascending Dosed of HSK31858 in Healthy Volunteers
Brief Title: A Study of Safety, Tolerability, and Pharmacokinetics of Single Ascending Dosed of HSK31858 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Haisco Pharmaceutical(Australia) Pty Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSK31858-101
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: HSK31858; NCFBE; health; phase I
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK31858, single dose (Experimental): 5 cohorts with single doses starting with 5 mg HSK31858 as tablet.
  Interventions: Drug: HSK31858, tablet
- Placebe, single dose (Placebo Comparator): 5 cohorts with matching placebo to HSK31858 as tablet.
  Interventions: Drug: Placebo, tablet

INTERVENTIONS:
Drug: HSK31858, tablet — Starting dose in single ascending dose: 5 mg
  Arms: HSK31858, single dose
Drug: Placebo, tablet — Matching placebo
  Arms: Placebe, single dose

SUMMARY:
This is a Phase I, single-dose escalation clinical trial for HSK31858 conducted in healthy volunteers. The safety, tolerability, and pharmacokinetics of HSK31858 tablet in healthy volunteers will be evaluated using a randomized, double-blind, placebo-controlled trial design.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at Screening.
3. Body mass index ≥ 18.0 and ≤ 30.0 kg/m2, with a body weight ≥ 50 kg at Screening.
4. Be nonsmokers (including tobacco, e-cigarettes, and marijuana) for at least 1 month prior to first study drug administration.
5. Medically healthy without clinically significant abnormalities at Screening and predose on Day 1, including:

   1. Physical examination without any clinically relevant findings.
   2. Systolic blood pressure in the range of 90 to 140 mmHg and diastolic blood pressure in the range of 50 to 90 mmHg after 5 minutes in supine position.
   3. Heart rate in the range of 50 to 100 bpm after 5 minutes rest in supine position.
   4. Body temperature, between 35.0°C and 37.7°C.
   5. No clinically significant findings in serum chemistry, hematology, coagulation, and urinalysis tests as deemed by the Investigator.
6. Conventional 12-lead ECG recording in triplicate (the mean of triplicate measurements will be used to determine eligibility at Screening and predose on Day 1) consistent with normal cardiac conduction and function, including:

   * Normal sinus rhythm with HR between 50 and 100 bpm, inclusive.
   * QT interval corrected using the Fridericia method (QTcF) between 350 to 450 msec for male subjects and 350 to 470 msec for female subjects, inclusive.
   * QRS duration of < 120 msec.
   * PR interval of ≤ 210 msec.
   * Electrocardiogram morphology consistent with healthy cardiac ventricular conduction and normal rhythm, and with measurement of the QT interval.
   * No family history of short or long QT syndrome.
   * No history of risk factors for torsade de pointes or the diagnosis.
7. Women of childbearing potential must be non-pregnant and non-lactating, and must use an acceptable, highly effective double contraception from Screening until at least 30 days after last dose, including the Follow-up period. Double contraception is defined as a condom AND one other form of the following:

   * Established hormonal contraception (OCPs, long-acting implantable hormones, injectable hormones).
   * A vaginal ring or an IUD.
   * Documented evidence of surgical sterilization at least 6 months prior to Screening (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post-vasectomy documentation of the absence of sperm in semen] provided the male partner is a sole partner).

   Women not of childbearing potential must be postmenopausal for ≥12 months. Postmenopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrhoeic female subjects. Females who are abstinent from heterosexual intercourse will also be eligible.

   Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not considered highly effective methods of birth control. Subject complete abstinence for the duration of the study and for 1 month after the last study treatment is acceptable.

   Female subjects who are in same sex relationships are not required to use contraception.

   WOCBP must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study.
8. Male subjects must be surgically sterile (> 30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, the subject and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from Screening until study completion, including the Follow-up period. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring, or an IUD. Subjects with same sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle. Males must not donate sperm for at least 90 Days after the last dose of study drug.
9. Have suitable venous access for blood sampling.
10. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.
11. Subjects must have no relevant dietary restrictions and be willing to consume standard meals provided during the confinement period.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by the PI to be clinically relevant.
2. A primary diagnosis of chronic obstructive pulmonary disease or asthma as deemed by Investigator.
3. Subjects has increased risk of infection:

   1. History and/or presence of tuberculosis (TB).
   2. Body temperature of > 37.7℃.
   3. Blood neutrophil count <1.7 × 109/L, or white blood cell count < 4.0×109/L (Screening and Day -1).
   4. Is in high risk-group (i.e., men who have had unprotected sex with men, women who have had sex without a condom with men who have sex with men, people who have had sex without a condom with a person who has lived or travelled in Africa, people who inject drugs, people who have had sex without a condom with somebody who has injected drugs, people who have caught another sexually transmitted infection, people who have received a blood transfusion while in Africa, eastern Europe, the countries of the former Soviet Union, Asia or central and southern America) for human immunodeficiency virus (HIV) infection within the last 6 months.
   5. Other latent or chronic infections (e.g., recurrent sinusitis, genital or ocular herpes, urinary tract infection) or at risk of infection (surgery, trauma, or significant infection) within 3 months of Screening, or history of skin abscesses within 3 months of Screening.
   6. Clinically significant lower respiratory tract infection not resolved within 4weeks prior to Screening, as determined by the PI.
   7. Volunteers with active malignancy or neoplastic disease in the previous 5 years other than superficial basal cell carcinoma.
   8. Disease history suggesting abnormal immune function or use of or plans to use systemic immunosuppressive (e.g., corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) during the study or within 4 months prior to the first study drug administration.
   9. Volunteers who have received live or live-attenuated vaccine in the 4 weeks prior to dosing.
   10. High-sensitivity C-reactive protein > upper limit of normal (ULN) at Screening and on Day -1.
4. Some subjects lacking functional Dipeptidyl peptidase 1 (DPP1) enzyme have been described to have periodontitis and palmoplantar hyperkeratosis:

   1. Subjects with signs of current gingivitis/periodontitis. Gingival evaluation (by inspection) will be performed by a dental hygienist or trained study physician.
   2. Subjects with a history of hyperkeratosis or erythema in palms or soles.
5. Liver function test results (i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT], and gamma glutamyl transferase [GGT]) and total bilirubin elevated more than 1.2 fold above the ULN.
6. Positive test results for active HIV, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies (Abs).
7. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
8. Estimated creatinine clearance (CrCl) < 60 mL/min using the Cockcroft-Gault formula or serum creatinine more than 1.5-fold above the ULN.
9. History of alcohol abuse within 12 months prior to first study drug administration or positive alcohol breath test. Regular alcohol consumption defined as > 21 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit or a 125 mL glass of wine). Subject is unwilling to abstain from alcohol beginning 48 hours prior to admission to the CRU and during the confinement period.
10. History of substance abuse within 12 months prior to first study drug administration or positive drug test results. Subjects with a positive toxicology Screening panel (urine test including qualitative identification of barbiturates, THC, amphetamines, benzodiazepines, opiates, and cocaine).
11. Use of any prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 14 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, except occasional use of paracetamol. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest).
12. Demonstrated clinically significant (required intervention e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial.
13. Known hypersensitivity to any of the study drug ingredients.
14. For women of childbearing potential, a positive serum pregnancy test at Screening or a positive urine pregnancy test with confirmatory serum pregnancy test on Day -1.
15. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of first study drug administration.
16. Participation in another investigational clinical trial within 60 days prior to the first study drug administration and participation in more than 4 investigational drug studies within 1 year prior to Screening.
17. Any other condition or prior therapy that in the opinion of the PI would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.
18. Is an employee of an Investigator or Sponsor or an immediate relative of an Investigator.
19. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the Follow-up period.
20. History of life-threatening infection (e.g., meningitis).
21. Infections requiring parenteral antibiotics within the 6 months prior to Screening.
22. Healthy volunteers with tattoos.
23. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest) or participation in more than 4 investigational drug studies within 1 year prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | 7 days after dosing
  To assess the safety and tolerability of single oral dose of HSK31858 in healthy adult volunteers

SECONDARY OUTCOMES:
Cmax | within 15 minutes before administration until 72 hours after administration
  Maximum concentration
Tmax | within 15 minutes before administration until 72 hours after administration
  Time to maximum concentration
AUC0-last | within 15 minutes before administration until until 72 hours after administration
  Area under the drug concentration-time curve, from time 0h to 72h
t½ | within 15 minutes before administration until 72 hours after administration
  Apparent terminal half-life
CL/F | within 15 minutes before administration until 72 hours after administration
  Apparent total clearance of drug
Vd/F | within 15 minutes before administration until 72 hours after administration
  Apparent volume of distribution after oral administration

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gonen, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No